CLINICAL TRIAL: NCT00629512
Title: A Comparative Efficacy and Safety Study of Nexium (Esomeprazole Magnesium) Delayed-Release Capsules (40mg qd and 20mg qd) Versus Placebo for the Prevention of Gastric Ulcers Associated With Daily NSAID Use in Patients at Risk
Brief Title: Prevention of Gastric Ulcers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SH-NEN-0013
Record Dates: First submitted 2008-02-27; First posted 2008-03-06 (Estimated); Last update posted 2009-03-13 (Estimated); Status verified 2009-03

CONDITIONS: NSAID Associated Gastric Ulcers
Keywords: NSAID, Nexium, esomeprazole, Gastric Ulcers
MeSH Terms: conditions — Stomach Ulcer | interventions — Esomeprazole

ARMS (3):
- 1 (Experimental): 20mg oral daily
  Interventions: Drug: Esomeprazole
- 2 (Experimental): 40mg oral daily
  Interventions: Drug: Esomeprazole
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Esomeprazole — 20mg oral daily
  Other Names: Nexium
  Arms: 1
Drug: Esomeprazole — 40mg oral daily
  Other Names: Nexium
  Arms: 2
Drug: Placebo
  Arms: 3

SUMMARY:
Nonsteroidal anti-inflammatory drugs (NSAIDS) are often associated with gastric ulcers. This study looks at the prevention of these gastric ulcers with one of the three following treatment groups for up to 8 weeks: esomeprazole 40 mg once daily; esomeprazole 20 mg once daily; versus placebo; in patients at risk.

ELIGIBILITY:
Inclusion Criteria:

1. No gastric or duodenal ulcer on baseline endoscopy.
2. A clinical diagnosis of a chronic condition that requires daily NSAID treatment for at least 6 months.
3. Other inclusion criteria, as defined in the protocol.

Exclusion Criteria:

1. History of esophageal, gastric or duodenal surgery, except the simple closure of an ulcer.
2. History of severe liver disease, including (but not limited to) cirrhosis and acute or chronic hepatitis.
3. Other criteria, as defined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Estimated)
Dates: Start 2001-03; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of esomeprazole 40 mg qd versus placebo and esomeprazole 20 mg qd versus placebo for up to 6 months of the treatment for the prevention of gastric (and/or duodenal) ulcers in patients receiving daily NSAID therapy and being at risk | Assessments at Week 0, Week 4, Week 12, Week 26

SECONDARY OUTCOMES:
Investigator-assessed symptoms, defined as control of NSAID-associated GI symptoms for up to 6 months of treatment with esomeprazole 40 mg qd versus placebo and esomeprazole 20mg qd versus placebo in patients receiving daily NSAID therapy. | Assessments at Week 0, Week 4, Week 12, Week 26
Safety and tolerability of esomeprazole 40 mg qd versus placebo and esomeprazole 20mg qd versus placebo for up to 6 months of treatment in patients receiving daily NSAID therapy | Assessments at Week 0, Week 4, Week 12, Week 26

CONTACTS AND LOCATIONS:
Overall Officials: Professor Chris Hawkey, Principal Investigator — Queens Medical Centre; Paula Fernstrom, Study Director — Nexium Global Product Director, AstraZeneca